CLINICAL TRIAL: NCT01817569
Title: Specific Clinical Experience Investigation for Long-term Use of Exenatide (Byetta Subcutaneous Injection)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5550C00001; EUPAS19606 (Registry Identifier: ENCePP)
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus (DM); Byetta; Exenatide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Byetta

SUMMARY:
The purpose of this investigation is to describe general safety profile of type II Diabetes Mellitus (DM) Japanese patients under exenatide therapy in real world medical practices

DETAILED DESCRIPTION:
Specific Clinical Experience Investigation for long-term use of exenatide (Byetta subcutaneous injection).

ELIGIBILITY:
Inclusion Criteria:

- Patient diagnosed with Type 2 Diabetes Mellitus and who is naive patient with Byetta.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are eligible to be included in the study if they meet all of the following criteria:
  The patient who is diagnosed with Type 2 Diabetes Mellitus and who is naive patient with Byetta.
  The patient follows the PI of Byetta.
Sampling Method: Non-Probability Sample
Enrollment: 2948 (Actual)
Dates: Start 2011-02-13 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence. | 3 years
  Number of Adverse Drug Reactions

SECONDARY OUTCOMES:
Mean change of HbA1c. | 3 years
  Change value of HbA1c from baseline as mean / median / minimum / max.
Amount of change of total score of Diabetes Treatment Satisfaction Questionnaire (DTSQs). | 3 years
  The Diabetes Treatment Satisfaction Questionnaire (DTSQs) was designed to make the initial assessment of total diabetes treatment satisfaction, treatment satisfaction in specific areas, and perceived frequencies of hyperglycemia and hypoglycemia. Each of the 8 items are scored on a scale of 0-6 where 0= very dissatisfied and 6= very satisfied. The higher score, the greater satisfaction with the treatment.
Mean change in weight. | 3 years
Mean change in blood pressure. | 3 years.
Mean change in lipid metabolism. | 3 years
  Change value of lipid metabolism from baseline as mean / median / minimum / max.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca
Locations (46):
- Japan (46):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5550C00001&attachmentIdentifier=846e4155-9a58-400f-86e0-771d7a6d697a&fileName=D5550C00001_redacted_CSR_synopsis.PDF&versionIdentifier=